CLINICAL TRIAL: NCT03204695
Title: A Prospective, Multicenter, Non-randomized, Post-market Clinical Follow-up Study to Confirm Safety and Performance of the Coherex WaveCrest® Left Atrial Appendage Occlusion System in Patients With Non-valvular Atrial Fibrillation
Brief Title: WAVECREST Post Market Clinical Follow-Up (PMCF) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to device design modifications.
Sponsor: Coherex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHX_IP015
Record Dates: First submitted 2017-06-16; First posted 2017-07-02 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Atrial Fibrillation; Stroke; Left Atrial Appendage (LAA); LAA Closure; LAA Occlusion; WaveCrest
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- WaveCrest® (Experimental): Implant of WaveCrest® Left Atrial Appendage Occlusion System
  Interventions: Device: Percutaneous LAA Closure; Drug: Anticoagulation or Clopidogrel

INTERVENTIONS:
Device: Percutaneous LAA Closure — LAA Closure with the WaveCrest LAA Occlusion System (study device)
Drug: Anticoagulation or Clopidogrel — Subjects either continue on anticoagulation or receive clopidogrel

SUMMARY:
The WAVECREST PMCF Study is a prospective, non-randomized, multicenter study to confirm safety and performance of the Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System in the current medical practice setting in patients with non-valvular atrial fibrillation who are at increased risk for stroke. Up to 65 subjects may be enrolled at up to 15 study sites in Europe. Patients will be followed through 45 days post-procedure.

DETAILED DESCRIPTION:
The Coherex WaveCrest® Left Atrial Appendage Occlusion System is designed to permanently occlude the Left Atrial Appendage (LAA).

ELIGIBILITY:
The criteria for implant are in accordance to the current version of the Instructions for Use:

Inclusion Criteria:

1. Non-valvular paroxysmal, persistent, or permanent atrial fibrillation
2. 18 years of age or older
3. LAA anatomy amenable to treatment by percutaneous techniques
4. Risk factors for potential thrombus formation in the LAA
5. Willing to participate in the required follow-up visits and tests
6. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Ethics Committee or Institutional Review Board at the study site

Exclusion Criteria:

1. Known contraindication to percutaneous transseptal intervention
2. Left atrial appendage anatomy or size that will not allow appropriate implantation of the WaveCrest Implant
3. Intracardiac thrombus or other cardiac abnormality visualized prior to implant that would significantly impact procedural safety
4. Mitral valve stenosis < 1.5 cm2 or any stenosis consistent with rheumatic valvular disease or history of mitral valve replacement or repair
5. Known contraindication and/or allergy to nickel
6. Known active bacterial infection (i.e., sepsis, endocarditis)
7. Any known medical condition or overall health of the subject that could adversely affect procedural safety or potentially prevent the patient from completing all study required visits and tests.
8. Pregnant or breastfeeding women due to the risk of exposure to x-rays and medications associated with the implant procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom De Potter, MD, Principal Investigator — OLV Hospital
Locations (1):
- OLV Hospital, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Site-specific clinical study results may be published by Investigators in compliance with the Investigator Agreement and/or site agreement, as applicable.

RESULTS

PARTICIPANT FLOW:
Groups:
- Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System: In eligible participants, Coherex WaveCrest LAA occlusion system delivery sheath was used to deliver the implant percutaneously via the femoral vein through a transseptal puncture into the LAA.
Period: Overall Study
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
Started | 27
Treated: Intent-to-treat (ITT) Analysis Set | 24
Completed | 23
Not Completed | 4
Not completed — Death | 1
Not completed — Participant was treated with another device | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set consisted of all participants who signed the informed consent form, met all of the inclusion criteria and none of the exclusion criteria, and the Coherex Delivery sheath had been inserted into the participant's femoral vein.
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Mortality, Pericardial Effusion Requiring Intervention, Device Embolization (Major), Device Thrombus and Ischemic Stroke (Composite Primary Safety Endpoint)
Description: The primary safety outcome was the composite of death from any cause (all-cause mortality), pericardial effusion requiring intervention, device embolization (major), device thrombus and ischemic stroke up to 45 days. The analysis was based on Sponsor Assessment of Adverse Events data. Baseline was defined as the last available measurement on or before the date of the implantation procedure.
Time Frame: From baseline up to 45 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
Number analyzed (Participants) | 24
Participants
  All-cause mortality | 2
  Pericardial effusion requiring intervention | 2
  Device embolization (major) | 1
  Device thrombus | 0
  Ischemic stroke | 0

2. Secondary Outcome: Percentage of Participants Who Achieved Device Success
Description: Percentage of participants who achieved device success were reported. Device success was defined as the percentage of participants who had the device deployed and implanted in the correct position. Baseline was defined as the last available measurement on or before the date of the implantation procedure.
Time Frame: From baseline up to 45 days
Population: The ITT analysis set consisted of all participants who signed the informed consent form, met all of the inclusion criteria and none of the exclusion criteria, and the Coherex Delivery sheath had been inserted into the participant's femoral vein.
Measure: Number; unit: Percentage of Participants
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
Number analyzed (Participants) | 24
Percentage of Participants | 83.3

3. Secondary Outcome: Percentage of Participants Who Achieved Technical Success
Description: Percentage of participants who achieved technical success were reported. Technical success was defined as the percentage of participants who experienced successful placement and release of the occluder in the LAA with LAA closure (defined as no leak greater than [>]5 millimeters [mm] on color Doppler transesophageal echocardiogram [TEE]) and who were discharged from the cardiac catheterization laboratory without the occurrence of device-related complications. Baseline was defined as the last available measurement on or before the date of the implantation procedure.
Time Frame: From baseline up to 45 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
Number analyzed (Participants) | 24
Percentage of Participants | 79.2

4. Secondary Outcome: Percentage of Participants Who Achieved Procedural Success
Description: Percentage of participants who achieved procedural success were reported. Procedural success was defined as the percentage of participants who experienced successful placement and release of the occluder in the LAA with LAA closure (defined as no leak >5 mm on color Doppler TEE) and who were discharged from the cardiac catheterization laboratory without device-related complications and without procedure-related complications other than minor device embolization (defined as device embolization that can be resolved by percutaneous technique without surgical intervention or damage to surrounding cardiovascular structures). Baseline was defined as the last available measurement on or before the date of the implantation procedure.
Time Frame: From baseline up to 45 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
Number analyzed (Participants) | 24
Percentage of Participants | 75.0

ADVERSE EVENTS:
Time Frame: From baseline up to 45 days
Description: The intent-to-treat (ITT) analysis set consisted of all participants who signed the informed consent form, met all of the inclusion criteria and none of the exclusion criteria, and the Coherex Delivery sheath had been inserted into the participant's femoral vein. Baseline was defined as the last available measurement on or before the date of the implantation procedure.
Arm/Group | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System (N=24)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Device embolization (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System (N=24)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of this clinical study may be submitted for publication without regard for whether the trial results are positive or negative. Sponsor will be responsible for oversight of the publication process and will have oversight of publications of results of the trial, the Physician Advisory Committee may advise.

DOCUMENTS (2):
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03204695/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03204695/SAP_001.pdf